CLINICAL TRIAL: NCT00001612
Title: Long-Term Follow-Up of Patients Enrolled in the Early Treatment Diabetic Retinopathy Study (ETDRS)
Status: Completed | Type: Observational
Sponsor: National Eye Institute (NEI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970120; 97-EI-0120
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-05

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Long-Term Visual Outcome; Photocoagulation; J. H. Wilmer Eye Institute
MeSH Terms: conditions — Diabetic Retinopathy

SUMMARY:
Patients enrolled in the original Early Treatment Diabetic Retinopathy Study at the Clinical Center at Johns Hopkins Wilmer Eye Institute will be invited for a follow-up visit at the National Eye Institute. Visual function will be assessed with manifest refraction and standardized visual acuity measurement. The progression of retinopathy will be evaluated by ocular exam and fundus photography. A brief medical history will be obtained. The goal of this study is to evaluate the long-term results of patients whose diabetic retinopathy was treated with different strategies of scatter and/or focal laser photocoagulation.

DETAILED DESCRIPTION:
To evaluate the long-term clinical course and prognosis of diabetic retinopathy treated with different strategies of scatter and/or focal laser photocoagulation in patients enrolled in the Early Treatment Diabetic Retinopathy Study (ETDRS).

ELIGIBILITY:
Patient was originally enrolled in the Early Treatment Diabetic Retinopathy Study at the Johns Hopkins Wilmer Eye Institute.

Patient not previously enrolled are not eligible.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170
Dates: Start 1997-05; Study Completion 2000-08

CONTACTS AND LOCATIONS:
Locations (1):
- National Eye Institute (NEI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ferris FL 3rd. How effective are treatments for diabetic retinopathy? JAMA. 1993 Mar 10;269(10):1290-1. No abstract available. PMID 8437309